CLINICAL TRIAL: NCT01866007
Title: Phase 1, Open-label, Randomized, Parallel Study to Assess the Pharmacokinetic Comparability of 2 Formulations and to Evaluate Pharmacokinetic Comparability of Guselkumab (CNTO1959) Delivered by 2 Different Devices in Healthy Subjects
Brief Title: A Study to Assess the Pharmacokinetic Comparability of Guselkumab (CNTO1959) When Delivered by 2 Different Devices and as 2 Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100969; CNTO1959NAP1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: Healthy; Guselkumab; CNTO1959; Pharmacokinetics; UltraSafe Passive Delivery System (PFS-U); Prefilled syringe facilitated injection device (PFS FID)
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Group 1 (Experimental): 40 participants will receive a single subcutaneous (SC) injection of 100 mg guselkumab prepared from lyophilized formulation.
  Interventions: Drug: Guselkumab (lyophilized formulation)
- Group 2 (Experimental): 40 participants will receive a single SC injection of 100 mg guselkumab, liquid formulation with UltraSafe Passive Delivery System (PFS-U).
  Interventions: Drug: Guselkumab (liquid formulation with PFS-U)
- Group 3 (Experimental): 40 participants will receive a single SC injection of 100 mg guselkumab, liquid formulation with a prefilled syringe facilitated injection device (PFS FID).
  Interventions: Drug: Guselkumab (liquid formulation with PFS FID)
- Group 4 (Experimental): 20 participants will receive a single intravenous (IV) infusion of 100 mg guselkumab prepared from liquid formulation.
  Interventions: Drug: Guselkumab (liquid formulation)

INTERVENTIONS:
Drug: Guselkumab (lyophilized formulation) — Participants will receive a single SC injection of 100 mg guselkumab prepared from lyophilized formulation.
  Other Names: CNTO1959
  Arms: Group 1
Drug: Guselkumab (liquid formulation with PFS-U) — Participants will receive a single SC injection of 100 mg guselkumab, liquid formulation with PFS-U.
  Other Names: CNTO1959
  Arms: Group 2
Drug: Guselkumab (liquid formulation with PFS FID) — Participants will receive a single SC injection of 100 mg guselkumab, liquid formulation with PFS FID.
  Other Names: CNTO1959
  Arms: Group 3
Drug: Guselkumab (liquid formulation) — Participants will receive a single IV infusion of 100 mg guselkumab prepared from liquid formulation.
  Other Names: CNTO1959
  Arms: Group 4

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (what the body does to the medication) comparability of guselkumab in lyophilized and liquid formulations. Also to evaluate pharmacokinetic comparability of liquid formulation of guselkumab when delivered as prefilled syringe with UltraSafe Passive Delivery System [PFS-U] or with a prefilled syringe facilitated injection device [PFS FID]) following a single subcutaneous (SC) administration of 100 mg guselkumab in healthy participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), parallel study (each group of participants will be treated at the same time) of guselkumab in healthy participants. Approximately 140 participants will be randomly assigned in the ratio 2:2:2:1 in to 4 treatment groups: Group 1 (SC injection of lyophilized formulation), Group 2 (subcutaneous [SC] injection of liquid formulation with PFS-U), Group 3 (SC injection of liquid formulation with PFS-FID), and Group 4 (IV infusion of liquid formulation). The study consists of 3 phases: screening (up to 4 weeks), open-label treatment and inpatient follow up (1 week) and outpatient follow up (11 weeks). Safety evaluations will include assessment of adverse events, vital signs, physical examination, electrocardiograms, injection-site reactions, and clinical laboratory tests. The total duration of the study for each participant will be approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant with no clinically significant abnormalities
* Have a weight in the range of 60 kg to 90 kg for male participants; have a weight in the range of 50 kg to 80 kg for female participants
* Have a body mass index (BMI) of 18.5 kg/m2 to 29.0 kg/m2
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Participant has a history of any clinically significant medical illness including liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances, ophthalmological disorders, neoplastic disease, urinary tract diseases, or dermatological disease
* Currently have any known malignancy or have a history of malignancy
* Participant has a known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human proteins to monoclonal antibodies or antibody fragments
* Have had a Bacillus Calmette-Guérin (BCG) vaccination within 12 months of screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2013-05-09 (Actual); Primary Completion 2013-09-20 (Actual); Study Completion 2013-10-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) of guselkumab | Day 1 through Week 12
Area under the curve (AUC) from time 0 to 70 days of guselkumab | Day 1 through Week 12

SECONDARY OUTCOMES:
Absolute bioavailability of guselkumab | Day 1 through Week 12
  Bioavailability will be evaluated by using formula: AUC from time zero to infinity with extrapolation of the terminal phase of SC injection divided by AUC from time zero to infinity with extrapolation of the terminal phase of IV infusion of guselkumab and multiplied by 100.
Immunogenicity of guselkumab | Day 1 through Week 12
  Plasma levels of antibodies to guselkumab for evaluation of potential immunogenicity.
Number of participants with adverse events as a measure of safety and tolerability | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Tempe, Arizona
  - Lincoln, Nebraska
  - Neptune City, New Jersey

REFERENCES:
- See also: Phase 1, Open-label, Randomized, Parallel Study to Assess the Pharmacokinetic Comparability of 2 Formulations and to Evaluate Pharmacokinetic Comparability of Guselkumab (CNTO 1959) Delivered by 2 Different Devices in Healthy Subjects — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR100969&attachmentIdentifier=5e6af0a1-76da-4da5-9273-5f01fedffd68&fileName=CR100969_CSR_Synopsis.pdf&versionIdentifier=